CLINICAL TRIAL: NCT04284085
Title: Evaluation of a Psychoeducational Intervention for People With Suicidal Behaviour in the Penitentiary Environment. N'VIU Project
Acronym: N'VIU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Hospitalari de Vic (Other)
Collaborators: Government of Catalonia (Unknown)
Responsible Party: Principal Investigator, Dr. Pere Roura-Poch, Head of epidemiology, Consorci Hospitalari de Vic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AC277
Record Dates: First submitted 2020-02-17; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): There will be psycho-educational groups of 10 to 12 people, led by two professionals, one of them will always be a psychologist and an educator. In some sessions, other collaborators will be invited to participate, such as psychiatrists, educators, social workers, etc. who may act as external observers or implement the session. The number of sessions will be 13, one or two sessions a week and duration of 90 minutes.
  Interventions: Other: Psychoeducational intervention
- Control group (No Intervention): They will receive a fact sheet on suicide and also tips on how to increase suicidal ideation.

INTERVENTIONS:
Other: Psychoeducational intervention — Psycho-educational groups of 10 to 12 people, led by two professionals, one of them will always be a psychologist and an educator. In some sessions, other collaborators will be invited to participate, such as psychiatrists, educators, social workers, etc. who may act as external observers or implement the session. The number of sessions will be 13, one or two sessions a week and duration of 90 minutes.
  Arms: Intervention group

SUMMARY:
Objective. The main objective is to determine the effectiveness of a psychoeducational program conducted by rehabilitation professionals to reduce the number of suicidal behaviors in prisons.

Methodology. The design of the study will be a multicenter, randomized, two-group clinical trial with blind evaluation of response variables, one year follow-up. The study population will be a male and female prison population of a total of two Catalan prisons. As a dependent or outcome variable, the total number of suicidal behaviors recorded for 12 months after the intervention will be determined. As independent variables, socio-demographic, clinical and prison situation variables will be collected. The suicidal ideation will be measured with the Columbia-Suicide Severity Rating Scale (C-SSRS). The anxiety and depression with Hamilton scale for assessing anxiety (HDRS) and the Hamilton scale for assessing severity of depressive symptoms (HAM-D). The EuroQoL-5D Health Questionnaire (EQ-5D) to measure quality of life. And a satisfaction survey of psychoeducational group intervention. Participants who meet the inclusion criteria will be divided into two groups, an intervention group that will conduct group sessions with a frequency of two per week and duration of 90 minutes for a total of 13 sessions, and a control group that will receive information on suicide counseling.

Discussion. Mortality from suicide is higher in the prison population than in the general population. This project aims to evaluate the effect of a psychoeducational intervention on reducing the number of suicidal behaviors in prison, in order to evaluate their implementation at the level of the entire prison network.

ELIGIBILITY:
Inclusion Criteria:

-People who have attempted suicide or a risk of suicide moderate to high.

Exclusion Criteria:

* People with a mental disorder in a state of acute exacerbation
* Intellectual disability
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-02-17 (Actual)

PRIMARY OUTCOMES:
Number of suicidal behaviours | 12 months
  Total number of suicidal behaviors recorded during 12 months after the start of the study in both groups.

SECONDARY OUTCOMES:
Severity of suicidal ideation | 6 months
  Severity of suicidal ideation (Columbia-Suicide Severity Rating Scale, C-SSRS). Intensity of Ideation subscale, the total score ranges from 2 to 25,with a higher number indicating more intense ideation and greater risk.
Levels of Anxiety | 6 months
  Hamilton Anxiety Rating Scale (HARS): Total score range of 0-56, where <17 indi-cates mild severity, 18-24 mild to moderate severity and25-30 moderate to severe.
Levels of depression | 6 months
  Hamilton Depression Rating Scale (HDRS). Score: 0-7: No depression; 8-13: Mild depression; 14-18: Moderate depression; 19-22: Severe depression and ≥ 23: Very severe depression.
Level of Quality of life: EuroQoL-5D Health Questionnaire, EQ-5D | 6 months
  Quality of life (EuroQoL-5D Health Questionnaire, EQ-5D). Score: 0 (worst imagined state of health) to 100 (best imagined state of health).

CONTACTS AND LOCATIONS:
Locations (1):
- Vic University Hospital, Vic, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617